CLINICAL TRIAL: NCT07322198
Title: Effects of Gong's Mobilization With and Without Scapular High Lift on Shoulder Range of Motion and Functional Recovery in Adhesive Capsulitis; a Randomized Clinical Trial
Brief Title: Effects of Gong's Mobilization With and Without Scapular High Lift on Shoulder Range of Motion and Functional Recovery in Adhesive Capsulitis.
Acronym: Gongs Mob
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Management and Technology Sialkot Pakistan (Other)
Responsible Party: Principal Investigator, Danyal Ahmad, Head Of Department (HOD), University of Management and Technology Sialkot Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: kuhs/dpt/umt-skt-027
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Adhesive Capsulitis
Keywords: adhesive capsulitis; shoulder; capsulitis; gongs mobilization; scapular high-lift
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A (GONG'S MOBILIZATION WITH SCAPULAR HIGHLIFTS) (Experimental): GROUP A (GONG'S MOBILIZATION WITH SCAPULAR HIGHLIFTS) containing 21 participants who will be given Gong's mobilization with scapular high lifts for 30 minutes along with the conventional physiotherapy.
  Interventions: Other: Experimental: GROUP A (GONG'S MOBILIZATION WITH SCAPULAR HIGHLIFTS)
- GROUP B (GONG'S MOBILIZATION WITHOUT SCAPULAR HIGHLIFTS) (Experimental): GROUP B (GONG'S MOBILIZATION WITHOUT SCAPULAR HIGHLIFTS) containing 21 participants who were given Gong's mobilization without scapular high lifts for 30 minutes along with the conventional physiotherapy
  Interventions: Other: Experimental: GROUP B (GONG'S MOBILIZATION WITHOUT SCAPULAR HIGHLIFTS)

INTERVENTIONS:
Other: Experimental: GROUP A (GONG'S MOBILIZATION WITH SCAPULAR HIGHLIFTS) — In this technique, the therapist applies a sustained lateral glide to the humeral head while the patient actively performs shoulder elevation or abduction. Scapular high lifting is encouraged during the movement to assist shoulder elevation. The technique is performed within a pain-free range to reduce pain and improve shoulder mobility and functional movement.
  Arms: GROUP A (GONG'S MOBILIZATION WITH SCAPULAR HIGHLIFTS)
Other: Experimental: GROUP B (GONG'S MOBILIZATION WITHOUT SCAPULAR HIGHLIFTS) — Patients received Gong's mobilization without allowing scapular high lifting. The therapist applied a lateral glide to the humeral head while the patient performed pain-free shoulder elevation or abduction. Scapular movement was controlled to avoid compensation, aiming to reduce pain and improve shoulder mobility and function.
  Arms: GROUP B (GONG'S MOBILIZATION WITHOUT SCAPULAR HIGHLIFTS)

SUMMARY:
This study aims to compare the effectiveness of Gongs Mobilization with and without scapular High-lift in the management of Adhesive Capsulitis, focusing on specific outcomes like pain, functional outcomes, and work productivity.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial with a sample size of 42 participants, as calculated by the G power tool, with 5 % attrition rate, diagnosed with Adhesive Capsulitis. Subjects will be selected through non-probability convenient sampling based on inclusion and exclusion criteria, and randomly assigned into two groups, with 21 participants in each group. Group A will receive Gong mobilization with scapular high-lift, while Group B will receive Gong mobilization without scapular high-lift, both in conjunction with conventional therapy. Demographic Data will also be collected. Baseline and post-intervention data will be collected using SPADI, NPRS, and a goniometer. Data will be analyzed by using IBM SPSS 26.0. At the same time, the Shapiro-Wilk test will be applied to check normality.

ELIGIBILITY:
Inclusion Criteria:

* Participants, including both males and females.
* aged 40 to 60 years.
* Diagnosed with unilateral Adhesive capsulitis at the 2nd or 3rd stage of the disease

Exclusion Criteria:

* History of any trauma, tumor, fracture, surgery, or infection in a shoulder joint.
* Patient with pregnancy and a history of abnormal neurological status (radiculopathy, stroke with hemiplegia, brachial plexus injury).
* Restricted shoulder due to burns or postoperative scars.
* Moderate or High levels of diabetes.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
NUMERICAL PAIN RATING SCALE (NPRS) | 4 Weeks
  It is a fundamental tool used to evaluate pain intensity and pain tolerance. Subjects can rate their pain from 0 (no pain at all) to 10 (pain as bad as it could be) to check whether the pain is acute or chronic. 42. The test-retest reliability coefficient, the intra-class correlation coefficient (ICC) for NPRS, is 0.74, and the minimal clinically important difference (MCID) is 1.1 points

SECONDARY OUTCOMES:
SHOULDER PAIN AND DISABILITY INDEX (SPADI) | 4 Weeks
  SPADI is used to assess shoulder discomfort and impairment in patients with shoulder disorders. It consists of 13 items divided into two domains; a sub-scale that measures pain contains 5 items, and the other sub-scale consists of 8 items to assess disability. Every sub-scale has a scoring method that calculates the average (mean) at the end to make a score out of 100. A high score indicates greater impairment or disability, and vice versa. The reliability coefficient, the intra-class correlation, is ≥ 0.89, and its minimal clinically important difference (MCID) is 8 points
UNIVERSAL GONIOMETERY: | 4 Weeks
  The primary movements of the shoulder include flexion and extension, abduction and adduction, horizontal abduction and adduction, as well as lateral and medial rotation. While these movements are assessed at the glenohumeral joint, they rely on coordinated mobility at the sternoclavicular, acromioclavicular, and scapulothoracic joints41. For shoulder AROM, the reliability coefficient, intra-class correlation (ICC), is 0.53-0.6544. The ICC for PROM ranges from 0.87 to 0.99

CONTACTS AND LOCATIONS:
Overall Officials: HAMZA ZAHID, MS OMPT, Principal Investigator — University of Management and Technology Sialkot Pakistan
Locations (3):
- Pakistan (3):
  - Bethania Hospital Sialkot, Sialkot, Punjab Province
  - Raheem Surgical Hospital Sambrial, Sialkot, Punjab Province
  - University of Management and technology Sialkot Campus, Sialkot, Punjab Province

IPD SHARING:
Plan to Share IPD: Undecided
IPD may not be shared due to concerns regarding patient confidentiality, data ownership, ethical approvals, and consent limitations, as well as institutional or legal restrictions. Additionally, data may be withheld to protect ongoing analyses or unpublished results, or because the data contain sensitive information that cannot be fully anonymized.

REFERENCES:
- [Result] Challey T, Dutta2 A, Kalita A, Pyngrope4 HR. Effectiveness of Gong's Mobilization Over Myofascial Release Technique in Patients with Adhesive Capsulitis.: Life Sciences-Physiotherapy. International Journal of Life Science and Pharma Research. 2023 May 1;L134-44.
- [Result] Eldridge A, Lohman E, Asavasopon S, Gharibvand L, Michener L. External handheld loads affect scapular elevation and upward rotation during shoulder elevation tasks. Int Biomech. 2024 Dec;11(1):1-8. doi: 10.1080/23335432.2024.2332212. Epub 2024 Mar 19. Erratum In: Int Biomech. 2024 Dec;11(1):xx. doi: 10.1080/23335432.2025.2569220. PMID 38501436
- [Result] Poulose R, Navya T.V, Pawani DJ. A STUDY ON EFFECTIVENESS OF SCAPULAR PNF TECHNIQUES ON PAIN AND DYNAMIC STABILITY OF SCAPULA IN ADHESIVE CAPSULITIS OF SHOULDER JOINT. IJMAES. 2025;11(01):2271-86.